CLINICAL TRIAL: NCT05083663
Title: Effectiveness of Hyaluronidase as an Adjuvant to Bupivacaine in Ultrasound Guided Supraclavicular Brachial Plexus Block for Upper Limb Surgery
Brief Title: Effectiveness of Adding Hyaluronidase to Bupivacaine in Ultrasound Guided Supraclavicular Brachial Plexus Block
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hitham Mohammed Aly Elsayed, lecturer of anesthesia and surgical ICU, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Soh-Med-21.09.04
Record Dates: First submitted 2021-10-05; First posted 2021-10-19 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Pain
Keywords: hyaluronidase; supraclavicular block; buivacaine; ultrasound
MeSH Terms: conditions — Pain, Postoperative | interventions — Hyaluronoglucosaminidase

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): received bupivacaine 0.375 % 15 mL + normal saline 4ml +hyaluronidase 800 IU in 1 ml.
  Interventions: Drug: Hyaluronidase
- Group II (No Intervention): received bupivacaine 0.375% 15 mL + normal saline5 ml.

INTERVENTIONS:
Drug: Hyaluronidase — using hyaluronidase as an additive to bupivacaine
  Arms: Group I

SUMMARY:
Background Brachial plexus block is a good choice for surgeries of the upper limb because it provides good quality of anesthesia and analgesia especially in patients with multiple comorbidities and in ambulatory surgery. Hyalaluronidase is a local anesthetic adjuvant used for ophthalmologic surgery. We evaluated the effect of adding hyaluronidase to bupivacaine as regard the onset and duration of motor and sensory block in ultrasound guided supraclavicular brachial plexus block.

Methodology prospective, randomized and double-blind study conducted at Sohag University Hospital. A total of 40 adults scheduled for upper limb surgery, ASA I or II were randomly assigned into two groups (n=20). Group I received bupivacaine 0.375 % 15 mL + normal saline 4ml +hyaluronidase 800 IUin 1 ml. Group II received bupivacaine 0.375% 15 mL + normal saline5 ml. Both groups will be compared for onset and duration of sensory and motor block, duration of analgesia and complications.

Results The onset of sensory and motor block was significantly faster in hyaluronidase group than control group. Significant difference could not be detected in either duration of the sensory or motor block between the two groups.

Conclusion The use of hyaluronidase as an additive to bupivacaine fastens the onset of sensory and motor block of the brachial plexus in supraclavicular approach without affecting the duration of the block.

DETAILED DESCRIPTION:
This prospective, randomized, controlled and double-blind study was conducted at Sohag University Hospital after approval from institution review board and obtaining written informed consents from all participants. Forty participants, aged 18 to 60 years, American Society of Anesthesiologists class I and II, scheduled for elective surgery of the upper extremities were included in this study. Participants who refuse or have allergy to local anesthetic or hyaluronidase or suffering from severe renal, hepatic, pulmonary, cardiac, neurologic, psychiatric or neuromuscular disease will be excluded from the study in addition to pregnant or lactating women, patients with morbid obesity, coagulation disorders as well.

Sealed envelopes technique was used to randomly assign patients to both study groups; Group I; received bupivacaine 0.375 % 15 mL + normal saline 4ml +hyaluronidase 800 IU in 1 ml.

Group II; received bupivacaine 0.375% 15 mL + normal saline5 ml. After arriving to the operative theater basic monitoring was applied and intravenous line was inserted. Midazolam 2mg and Fentanyl 50 mcg was administered intravenously to all participants 15 minutes before the procedure. Anesthesiologist who carried out the block and recorded the study measurements was blinded to the treatment groups.

The participants were in supine position with the head rotated to the opposite side and neck extended, 7 to 12 MHz linear ultrasound probe (SonoScape A5, SonoScape Co., Ltd., China) was placed above the clavicle to identify distal trunks or proximal divisions of the brachial plexus lateral and cephalad to the subclavian artery above the first rib. After ultrasound pre-scan and local infiltration with 3ml lidocaine 2%, 100 mm, 20 gauge nerve-stimulating needle (Locoplex®, VYGON, FRANCE) was inserted under real time ultrasound guided technique in line approach and advanced until reaching the brachial plexus sheath the needle was repositioned to allow local anesthetic spread around all trunks or divisions. Injection was stopped if an increased resistance to injection experienced or parathesia to avoid intra neural injection. All participants were transferred to post-anesthesia care unit postoperatively to be observed for the following measurements:

The primary measurement:

1. Onset of complete sensory block (time from injection to complete sensory block to pin prick).
2. Onset of complete motor block (time from injection to complete motor block).

Secondary measurements:

1. Duration of analgesia defined as time from injection to first analgesia request.
2. Duration of sensory block (time between injection and complete recovery of sensation)
3. Duration of motor block (time between injection and complete recovery of motor power)
4. Side effects and complications (hypotension, sedation, nausea vomiting, dry mouth, hematoma or pneumothorax, neuropathy) Participants were allowed to receive analgesia as ketorolac 30 mg intramuscularly as a rescue analgesia if VAS > 4.

Statistical analysis:

After performing the power analysis of the study , it is decided that each group should contain at least a minimum of 18 cases (90% power and 0.05%alpha error).Considering possible data loss due to technical reasons, each group was decided to be 20 patients.

Recorded data were subjected to statistical analysis using Statistical Package for Social Sciences (SPSS), Student's t-test was used for statistical analysis of demographic and hemodynamic data while unpaired t-test was applied for onset time and duration of sensory and motor blocks and was reconfirmed with the Wilcoxon W and Mann-Whitney U tests. Statistical significance was defined by P-value < 0.05. chi-square/Fischer's exact test was used for analysis of adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 60 years
* American Society of Anesthesiologists class I and II
* Scheduled for elective surgery of the upper extremities

Exclusion Criteria:

* allergy to local anesthetic or hyaluronidase
* Severe renal or hepatic disease
* Pulmonary, cardiac disease
* Neurologic, psychiatric disease
* Neuromuscular disease
* Pregnant or lactating women
* Morbid obesity
* Coagulation disorders as well

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Onset of complete sensory block | during the first 24 hours
  time from injection to complete sensory block to pin prick
Onset of complete motor block | during the first 24 hours
  time from injection to complete motor block

SECONDARY OUTCOMES:
duration of anlgesia | during the first 24 hours
  time from injection to first analgesia request
Duration of sensory block | during the first 24 hours
  time between injection and complete recovery of sensation
duration of motor block | during the first 24 hours
  time between injection and complete recovery of motor power
side effects | during the first 24 hours
  hypotension, sedation, nausea vomiting, dry mouth, hematoma or pneumothorax, neuropathy

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No